CLINICAL TRIAL: NCT00292162
Title: Radiofrequency Ablation for Atrial Fibrillation in Advanced Chronic Heart Failure
Brief Title: Curing Atrial Fibrillation in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Michael MacDonald, Cardiology ST6, NHS Greater Glasgow and Clyde
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/S0704/47
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Heart Failure; Atrial Fibrillation
Keywords: Chronic Heart Failure; Atrial Fibrillation; Radiofrequency Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation; Enalapril; Captopril; Perindopril; Lisinopril; Adrenergic beta-Antagonists; Metoprolol; Bisoprolol; Carvedilol

ARMS (2):
- medical therapy (Active Comparator): Standard therapy for heart failure with angiotensin converting enzyme inhibitors(ACE) - (Ramipril, enalapril, lisinopril, captopril, perindopril), beta-blocker (BB) - (carvedilol, bisoprolol, metoprolol), Aldosterone antagonists (spironolactone) +/- diuretics and digoxin
  Interventions: Drug: ACE inhibitor - ramipril, enalapril, captopril, perindopril, lisinopril; Drug: Beta Blocker (BB) - metoprolol, bisoprolol, carvedilol; Drug: Aldosterone Antagonists - spironolactone
- Radiofrequency ablation (RFA) (Active Comparator): Isolation of the pulmonary veins using radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: radiofrequency ablation — isolation of the pulmonary veins with radiofrequency ablation (RFA)
  Other Names: radiofrequency ablation (RFA); pulmonary vein isolation (PVI)
  Arms: Radiofrequency ablation (RFA)
Drug: ACE inhibitor - ramipril, enalapril, captopril, perindopril, lisinopril — Evidence based treatment for heart failure. Dose and type will depend on patient tolerability.
  Arms: medical therapy
Drug: Beta Blocker (BB) - metoprolol, bisoprolol, carvedilol — Evidence based treatment for heart failure. Dose and type will depend on patient tolerance.
  Arms: medical therapy
Drug: Aldosterone Antagonists - spironolactone — Evidence based treatment for heart failure. Dose and type will depend on patient to treatment.
  Arms: medical therapy

SUMMARY:
Heart failure is a condition that occurs when the heart muscle weakens and no longer contracts normally. Half of these patients have an irregularity of heart rhythm called atrial fibrillation (AF). Patients with both heart failure and AF spend more time in hospital, and die earlier than those with heart failure alone. AF is difficult to treat with conventional methods in patients with heart failure. Radiofrequency ablation is a new technique used to cure AF. The investigators aim to establish if radiofrequency ablation for atrial fibrillation in patients with advanced heart failure can result in marked improvement in the function of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Persistent atrial fibrillation (AF)
* New York Heart Association (NYHA) II, III and IV chronic heart failure (CHF) despite optimal medical therapy for at least 3 months
* left ventricular ejection fraction (LVEF) <35% - as measured by radionuclide ventriculography (RNVG)
* Patients with CHF secondary to ischaemic and non-ischaemic aetiology

Exclusion Criteria:

* QRS duration >150ms (or QRS 120-150 with evidence of mechanical cardiac dysynchrony)
* Magnetic resonance imaging (MRI) - incompatible metallic (ferrous) prosthesis
* Primary valvular disease as a cause of CHF
* Reversible causes of CHF
* Acute myocarditis
* Patients aged 18 or less
* Patients having undergone revascularisation procedures within 6 months
* Paroxysmal AF
* Pregnancy
* Expected cardiac transplantation within 6 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek T Connelly, MBChB, Principal Investigator — Glasgow Royal Infirmary
Locations (1):
- Glasgow Royal Infirmary, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] MacDonald MR, Connelly DT, Hawkins NM, Steedman T, Payne J, Shaw M, Denvir M, Bhagra S, Small S, Martin W, McMurray JJ, Petrie MC. Radiofrequency ablation for persistent atrial fibrillation in patients with advanced heart failure and severe left ventricular systolic dysfunction: a randomised controlled trial. Heart. 2011 May;97(9):740-7. doi: 10.1136/hrt.2010.207340. Epub 2010 Nov 4. PMID 21051458

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Therapy: This consisted of standard treatment of heart failure as per international guidelines. Treatment generally included use of ace-inhibitors (captopril, enalapril, lisinopril, perindopril, ramipril), beta blocker (metoprolol, carvedilol, bisoprolol) and aldosterone antagonists (spironolactone). Obviously actual combination dose and type of drug used dependent on patient comorbidity and tolerance.
- Radiofrequency Ablation: Patients underwent isolation of the pulmonary veins with radiofrequency ablation. This was performed a maximum of 2 times to try to acheive sinus rhythm. All patients also received background heart failure treatment as per international guidelines.
Period: Overall Study
Arm/Group | Medical Therapy | Radiofrequency Ablation
Started | 19 | 22
Completed | 18 | 20
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Therapy | Radiofrequency Ablation | Total
Number analyzed (Participants) | 19 | 22 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (8) | 62 (6.7) | 63 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular Ejection Fraction by Magnetic Resonance Imaging (MRI)%
Description: left ventricular ejection fraction (LVEF) is a measure of the % of blood ejected from the ventricle in one heart beat. It is a measure of cardiac function. We measured LVEF at baseline and at 6 months, to assess whether there had been a change in the patients cardiac function over time.
Time Frame: baseline and 6 months
Population: Number of patients analyzed is different from number of patients enrolled because some of the outcomes could not be measured in some patients ie the patient did not tolerate an mri or dropped out of the study
Measure: Mean (Standard Deviation); unit: percentage of blood ejected in one beat
Arm/Group | Medical Therapy | Radiofrequency Ablation
Number analyzed (Participants) | 19 | 19
percentage of blood ejected in one beat | 2.8 (6.8) | 4.5 (11.1)

2. Secondary Outcome: Plasma B-type Natriuretic Peptide (BNP)
Description: venous blood taken to assess levels of the above peptide. High evels of the peptide are associated with adverse prognosis. Blood levels are taken at baseline and 6 months. The change over 6 months is assessed, thereore it is possible to have a negative number if the level falls.
Time Frame: baseline and 6 months
Population: Number of patients analyzed is different from number of patients enrolled because some of the outcomes could not be measured in some patients ie the patient did not tolerate a blood test or dropped out of the study
Measure: Mean (Standard Deviation); unit: picograms per millilitre
Arm/Group | Medical Therapy | Radiofrequency Ablation
Number analyzed (Participants) | 18 | 20
picograms per millilitre | 85 (648) [-563 to 733] | -196 (1469) [-1665 to 1273]

3. Primary Outcome: Baseline Left Ventricular Ejection Fraction by Magnetic Resonance Imaging (MRI)
Description: Baseline Left Ventricular Ejection Fraction by Magnetic Resonance Imaging (MRI)in %
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of blood ejected in one beat
Arm/Group | Medical Therapy | Radiofrequency Ablation
Number analyzed (Participants) | 19 | 19
percentage of blood ejected in one beat | 43 (10) [33 to 53] | 36 (12) [24 to 48]

4. Primary Outcome: Left Ventricular Ejection Fraction by Magnetic Resonance Imaging (MRI)at 6 Months
Description: Left Ventricular Ejection Fraction as measured by Magnetic Resonance Imaging (MRI)at 6 months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of blood ejected in one beat
Arm/Group | Medical Therapy | Radiofrequency Ablation
Number analyzed (Participants) | 19 | 19
percentage of blood ejected in one beat | 46 (7) [39 to 53] | 41 (11) [30 to 52]

5. Secondary Outcome: Plasma B-type Natriuretic Peptide (BNP) at Baseline
Description: Plasma B-type Natriuretic Peptide (BNP) measured at basline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: picograms per millilitre
Arm/Group | Medical Therapy | Radiofrequency Ablation
Number analyzed (Participants) | 19 | 19
picograms per millilitre | 1846 (1687) [159 to 3533] | 2550 (2150) [400 to 4700]

6. Secondary Outcome: Plasma B-type Natriuretic Peptide (BNP) at 6 Months
Description: Plasma B-type Natriuretic Peptide (BNP)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: picograms per millilitre
Arm/Group | Medical Therapy | Radiofrequency Ablation
Number analyzed (Participants) | 19 | 19
picograms per millilitre | 1931 (1671) [260 to 3608] | 2354 (2632) [-278 to 4986]

ADVERSE EVENTS:
Arm/Group | Medical Therapy | Radiofrequency Ablation
Serious Adverse Events (participants affected / at risk) | 0/19 | 4/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Therapy (N=19) | Radiofrequency Ablation (N=22)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2)
heart failure hospitalisation (Cardiac disorders) | 0 (0) | 1 (1) — within 1 week of the procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No